CLINICAL TRIAL: NCT01464021
Title: A Post-Marketing Observational Study to Evaluate the Effectiveness of Adalimumab in Patients With Moderately to Severely Active Rheumatoid Arthritis in China
Status: Terminated | Type: Observational
Why Stopped: This study was prematurely terminated due to low enrollment
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-194
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-02

CONDITIONS: Arthritis; Rheumatoid
Keywords: Study; prospective; Rheumatoid; Observational study; Arthritis; Adalimumab
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab: Chinese adult participants with a diagnosis of rheumatoid arthritis (RA) (any disease duration) who meet the requirements per the local label for treatment with adalimumab. Participants must be naïve to adalimumab at the Baseline visit.

SUMMARY:
A post-marketing uncontrolled observational study to explore and describe the effectiveness of adalimumab, as prescribed according to the local product label, in patients with moderately to severely active rheumatoid arthritis (RA) in China.

DETAILED DESCRIPTION:
This post-marketing, multi-center, uncontrolled observational study will be conducted in an open-label, non-interventional setting, for RA patients using commercially available adalimumab administered subcutaneously (SC). Adalimumab effectiveness will be assessed based on data from clinic visits beginning at Baseline and continuing per standard of care for RA. The primary objective is to evaluate the effectiveness of adalimumab in improving patients' disease activity measured by Disease Activity Score (DAS28) at Week 12. The maximum observation period for each patient is approximately 52 weeks, as long as the patient continues to receive adalimumab injections. The study was terminated due to low enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient greater than or equal to 18 years of age with diagnosis of RA (Rheumatoid Arthritis) and no history of chronic arthritis before age 16.
2. Patient meets the requirements for treatment with adalimumab per the local product label.
3. Patient is naïve to adalimumab, and has not used any other immunomodulatory biologic* DMARD (Disease Modifying Antirheumatic Drugs) in the past 8 weeks before the Baseline visit (*rituximab may not have been used in the past 104 weeks before the Baseline visit).
4. Patient must be able and willing to provide written authorization (or informed consent where applicable) to disclose and use personal health information and comply with the requirements of this study protocol as well as agree to data being collected by Abbott.

Exclusion Criteria:

1. Patient is currently being treated with or has been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or five half lives (whichever is longer) of the drug prior to the Baseline visit.
2. Prior clinically active TB (tuberculosis): if patient has had prior clinically active TB, there should be documentation that a full course of appropriate anti-TB therapy was completed or an ongoing full course of appropriate anti-TB therapy has been started before initiation of adalimumab in accordance with the local product label; otherwise, the patient will not be eligible to participate in this study.
3. Patient who intends to take less than 6 consecutive (every other week) injections of adalimumab.
4. Patients should not be enrolled if they cannot be treated with adalimumab in accordance with the local product label or if the Investigator determines that they should not be enrolled based on his/her clinical judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adult participants with a diagnosis of rheumatoid arthritis (RA) (any disease duration) who meet the requirements per the local label for treatment with adalimumab. Participants must be naïve to adalimumab at the Baseline visit.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Carlson, Study Director — AbbVie
Locations (3):
- China (3):
  - Site Reference ID/Investigator# 64782, Guangzhou
  - Site Reference ID/Investigator# 65702, Shanghai
  - Site Reference ID/Investigator# 65706, Ürümqi

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab
Started | 26
Completed | 0
Not Completed | 26
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — various | 11

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least a Moderate European League Against Rheumatism (EULAR) Response
Description: A EULAR response reflects improvement in disease activity and attainment of a lower degree of disease activity based on the Disease Activity Score (DAS)28 score. The DAS28 score ranges from 0-10, with higher scores indicating more disease activity.
  A Good Response is defined as an improvement (decrease) in the DAS28 of more than 1.2 compared with Baseline and attainment of a DAS28 score of less than or equal to 3.2.
  A Moderate Response is defined as either:
  an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 from Baseline and attainment of a DAS28 score of less than or equal to 5.1 or, an improvement (decrease) in the DAS28 of more than 1.2 from Baseline and attainment of a DAS28 score of greater than 3.2.
  No Response is defined as either an improvement (decrease) in the DAS28 of less than or equal to 0.6, or an improvement (decrease) in the DAS28 of greater than 0.6 and less than or equal to 1.2 and attainment of a DAS28 of more than 5.1
Time Frame: Week 12
Population: Participants who received at least 6 consecutive injections of adalimumab (every other week) and have the necessary clinical data for both the Baseline and the Week 12 visit available.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 13
participants | 9

2. Secondary Outcome: Percent Change From Baseline in Disease Activity Score (DAS)28 Erythrocyte Sedimentation Rate (ESR)
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, erythrocyte sedimentation rate (ESR), and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score > 5.1 indicates high disease activity, ≤ 5.1 indicates moderate disease activity, ≤ 3.2 indicates low disease activity, and ≤ 2.6 indicates clinical remission.
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 15
percent change
  Week 4, n=15 | -34.2 (18.96)
  Week 8, n=12 | -38.0 (28.33)
  Week 12, n=13 | -42.4 (25.66)
  Week 26, n=3 | -62.4 (26.14)

3. Secondary Outcome: Percent Change From Baseline in Tender and Swollen Joint Counts
Description: Change in number of tender joints and swollen joints for 28 assessed joints.
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 19
Percent change
  Week 4 tender joint count, n=19 | -47.9 (38.64)
  Week 8 tender joint count, n= 14 | -44.4 (69.89)
  Week 12 tender joint count, n= 13 | -65.0 (42.89)
  Week 26 tender joint count, n= 4 | -93.8 (12.50)
  Week 4 swollen joint count, n=19 | -45.7 (39.33)
  Week 8 swollen joint count, n=14 | -43.9 (69.70)
  Week 12 swollen joint count, n=13 | -56.4 (55.75)
  Week 26 swollen joint count, n=4 | -96.9 (6.25)

4. Secondary Outcome: Percent Change From Baseline in C-reactive Protein
Description: C-reactive protein level in serum (mg/dL)
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 13
percent change
  Week 4, n=13 | 206.4 (808.73)
  Week 8, n=11 | -14.6 (91.82)
  Week 12, n=11 | 33.7 (175.17)
  Week 26, n=3 | -82.3 (29.23)

5. Secondary Outcome: Percent Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: Rate at which red blood cells sediment in a period of 1 hour, a non-specific measure of inflammation; a higher rate = more inflammation.
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 16
percent change
  Week 4, n=16 | -50.7 (29.60)
  Week 8, n=12 | -48.0 (35.77)
  Week 12, n=13 | -46.5 (42.14)
  Week 26, n=3 | -68.0 (35.91)

6. Secondary Outcome: Percent Change From Baseline in Patient's Global Assessment of Disease Activity
Description: A horizontal Visual Analog Scale (VAS) (100 mm) measure of the participant's global assessment of RA disease activity, where the participant was asked to place a vertical mark on the line to indicate how well their RA has been within the last 24 hours, ranging from 0 mm (very well) to 100 mm (very poorly).
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 19
percent change
  Week 4, n=19 | -44.8 (26.70)
  Week 8, n=14 | -55.5 (37.91)
  Week 12, n=13 | -55.8 (42.69)
  Week 26, n=4 | -66.0 (34.35)

7. Secondary Outcome: Percent Change From Baseline in Patient's Assessment of Pain
Description: A horizontal VAS (100 mm) measure of the participant's assessment of RA pain, where the participant was asked to place a vertical mark on the line to indicate how much pain they have had due to RA in the past week, ranging from 0 mm (no pain) to 100 mm (pain as bad as it could be).
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 19
percent change
  Week 4, n=19 | -48.8 (28.10)
  Week 8, n=14 | -57.9 (38.01)
  Week 12, n=13 | -54.1 (43.01)
  Week 26, n=4 | -67.2 (34.02)

8. Secondary Outcome: Percent Change From Baseline in Physician's Global Assessment of RA Disease Activity
Description: A horizontal VAS (100 mm) measure of the physician's global assessment of the participant's current RA disease activity, ranging from 0 mm (very good condition) to 100 mm (very bad condition).
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 19
percent change
  Week 4, n=19 | -45.7 (27.56)
  Week 8, n=14 | -55.9 (35.03)
  Week 12, n=13 | -53.3 (39.04)
  Week 26, n=4 | -63.4 (32.15)

9. Secondary Outcome: Percent Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI)
Description: The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3).
Time Frame: Weeks 4, 8, 12, 26
Population: Participants who received at least one injection of adalimumab and have the necessary clinical data available.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Adalimumab
Number analyzed (Participants) | 15
percent change
  Week 4, n=15 | -47.7 (47.24)
  Week 8, n=10 | -58.2 (45.53)
  Week 12, n=12 | -62.3 (42.27)
  Week 26, n=3 | -97.6 (4.12)

ADVERSE EVENTS:
Time Frame: From the time of signing of participant authorization or informed consent until 70 days following the last dose of study adalimumab.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=26)
Upper Respiratory Tract Infection (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment and high drop-out rate. Only serious adverse events and events leading to discontinuation were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.